CLINICAL TRIAL: NCT00563108
Title: A Double-blind Randomized Single-center Trial of Basiliximab for the Treatment of Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation.
Brief Title: Basiliximab for the Treatment of Acute Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Collaborators: Novartis Pharmaceuticals (Industry); The Hong Kong Blood Cancer Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 03-312 T312; HARECCTR0500037
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Graft vs Host Disease; Hematopoietic Stem Cell Transplantation
Keywords: Acute graft-versus-host disease post allogeneic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Basiliximab

INTERVENTIONS:
Drug: Basiliximab
Drug: Placebo

SUMMARY:
Graft-versus-host disease (GVHD) contributes substantially to transplant-related morbidity and mortality. Steroids remains first line therapy for acute GVHD but there is currently no consensus on second line therapy for those in whom steroids have been ineffective. Basiliximab has been shown to be a safe and effective immunosuppresant in the prevention and treatment of rejection after renal transplantation and its role in acute GVHD prophylaxis and treatment has been described favourably. This is a randomized control trial to investigate its efficacy and safety in the management of acute GVHD post allogeneic stem cell transplantation (SCT).

ELIGIBILITY:
Inclusion Criteria:

* Grade II to IV acute GVHD after SCT

Exclusion Criteria:

* Known allergy to basilixmab

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-06; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Resolution of GVHD by Day 12 | 12 days

SECONDARY OUTCOMES:
Duration and grading of acute GVHD | 100 days
Total dose of steroid and immunosuppresant | 100 days
Mortality, GVHD-related and all cause | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence SY Ma, Dr, Principal Investigator — Department of Medicine/ Haematology and Oncology, Queen Mary Hospital
Locations (1):
- The University of Hong Kong, Hong Kong, China